CLINICAL TRIAL: NCT00071422
Title: A Randomized, Double-blind, Placebo-controlled, Rising-dose, Multicenter Study to Evaluate the Efficacy and Safety of 90 Days of 300 or 600 mg Daily Subcutaneous Injections of INGAP Peptide in Insulin-using Type 2 Diabetes Mellitus Patients
Brief Title: Safety and Efficacy of INGAP-Peptide in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exsulin Corporation (Industry)
Responsible Party: Muhammad Rehman, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003069
Record Dates: First submitted 2003-10-22; First posted 2003-10-23 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — INGAP peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- placebo (Placebo Comparator): 1.5 mL SC injection, once daily for 90 days
  Interventions: Drug: placebo
- 300 mg INGAP Peptide (Experimental): 1.5 mL SC injection, once daily for 90 days
  Interventions: Drug: INGAP-Peptide
- 600 mg INGAP Peptide (Experimental): 1.5 mL SC injection, once daily for 90 days
  Interventions: Drug: INGAP-Peptide

INTERVENTIONS:
Drug: INGAP-Peptide — 1.5 mL, once daily, self-administered SC injection for 90 days
  Arms: 300 mg INGAP Peptide
Drug: INGAP-Peptide — 1.5 mL, once daily, self-administered SC injection for 90 days
  Arms: 600 mg INGAP Peptide
Drug: placebo — 1.5 mL, once daily, self-administered SC injection for 90 days
  Arms: placebo

SUMMARY:
Insulin is a chemical that the body needs in order to use or store sugar. It is made by a type of cell called a beta cell which resides in an organ known as the pancreas. Type 2 diabetes is a disease where the beta cells are unable to meet a person's insulin needs. Sugar levels rise in the blood as a result. INGAP-Peptide is being tested to attempt to create new beta cells in the pancreas, and to improve the ability to produce insulin in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria

* Age 35-70
* Using >20 Units of insulin per day
* HbA1c from 6.5% to 10%
* No islet antibodies
* Otherwise healthy

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2003-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Diabetes and Endocrine Associates, La Jolla, California
  - VA Hospital UCSD, San Diego, California
  - Diablo Clinical Research, Walnut Creek, California
  - Denver, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - MedStar Clinical Research Center, Washington D.C., District of Columbia
  - Future Care Studies, Springfield, Massachusetts
  - Mercury Street Medical, Butte, Montana
  - Diabetes-Endocrinology Center of WNY, Buffalo, New York
  - UNC Diabetes Care Center, Durham, North Carolina
  - Piedmont Medical Group, Winston-Salem, North Carolina
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Mountain View Clinical Research, Greer, South Carolina
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - University of Texas Health Science Center - Texas Diabetes Institute, San Antonio, Texas
  - DGD Research Associates, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia